CLINICAL TRIAL: NCT04029857
Title: Nutritional Supplementation for Esophageal Cancer Patients Undergoing Trimodality Therapy
Brief Title: Nutritional Supplementation in Reducing Complications in Patients With Locally Advanced Esophageal Cancer Undergoing Chemotherapy, Radiation Therapy, and/or Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0772; NCI-2019-04165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0772 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage III Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Esophageal Squamous Cell Carcinoma AJCC v8; Resectable Mass
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (standard of care) (Active Comparator): Patients receive standard of care nutritional supplementation.
  Interventions: Dietary Supplement: Nutritional Supplement Drink
- Group II (Impact Advanced Recovery) (Experimental): Patients receive Impact Advanced Recovery PO or via feeding tube BID on days 1-7 for weeks 1, 3, and 5 during chemotherapy and radiation therapy before surgery. Starting 5-7 days before surgery, patients receive Impact Advanced Recovery PO TID until surgery. Within 2 days following surgery, patients may continue to receive Impact Advanced Recovery via feeding tube at the discretion of the treating physician.
  Interventions: Dietary Supplement: Nutritional Supplementation

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement Drink — Given standard of care nutritional supplementation
  Other Names: Boost; Ensure; polymeric enteral nutrition formula
  Arms: Group I (standard of care)
Dietary Supplement: Nutritional Supplementation — Given Impact Advanced Recovery PO or via feeding tube
  Other Names: Supplementation
  Arms: Group II (Impact Advanced Recovery)

SUMMARY:
This phase III trial studies nutritional supplementation with Impact Advanced Recovery to see how well it works compared with standard nutritional supplementation in reducing complications in patients with esophageal cancer that has spread to nearby tissue or lymph nodes (locally advanced) who are undergoing chemotherapy, radiation therapy, and/or surgery. Impact Advanced Recovery may help to reduce the number of surgical complications, reduce toxicity, improve nutritional status before surgery, and reduce morbidity after surgery in patients with esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. When compared to the current standard of ad hoc nutritional supplementation on an as-needed basis, scheduled enteral supplementation with Impact Advanced Recovery during the course of neoadjuvant therapy (for those in the planned trimodality group), preoperatively, and postoperatively will improve patient wellbeing by reducing weight loss (measured at baseline, preoperatively, and at postoperative follow-up) incurred during the course of therapy and will permit maintenance of patient performance status.

SECONDARY OBJECTIVES:

I. Decrease rates of a composite outcome that includes anastomotic leaks, ileus, major pulmonary events (pneumonia, reintubation, tracheostomy), wound infection, postoperative mortality, chyle leaks, and other postoperative complications.

II. Improve overall survival. III. Return to pre-surgical activity level (measured by Eastern Cooperative Oncology Group [ECOG] at baseline, preoperatively, and at postoperative follow-up).

IV. Decrease postoperative length of stay. V. Decrease incidence of esophagitis during and after radiation therapy. VI. Improve rates of completion of all planned neoadjuvant therapies (defined as receipt of a minimum of 41.4 Gray and two cycles of chemotherapy).

VII. Improve rates of lymphopenia.

EXPLORATORY OBJECTIVES:

I. Maintain or improve serum levels of arginine, citrulline, and albumin, while maintaining or decreasing serum levels of asymmetric dimethylarginine (ADMA) and C-reactive protein.

II. Improve immune function using peripheral markers such as CD4 count, CD4:CD8 ratio, CD3 zeta, myeloid-derived suppressor cells (MDSCs), IL-6 (interleukin 6), and IL-7.

III. Increase densities of tumor-associated immune cells (TAICs; including CD3+, CD8+, CD45RO+, CD57+, CD4+, FOXP3+, granzyme B+, CD68+, PD1+ cells) within the tumor tissue.

IV. Reduce platelet-to-lymphocyte, monocyte-to-lymphocyte, and neutrophil-to-lymphocyte ratios as measured by routine clinical complete blood counts.

V. Composition of intratumoral, peritumoral, and enteric microbiome.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive standard of care nutritional supplementation.

GROUP II: Patients receive Impact Advanced Recovery PO or via feeding tube twice daily (BID) on days 1-7 for weeks 1, 3, and 5 during chemotherapy and radiation therapy before surgery. Starting 5-7 days before surgery, patients receive Impact Advanced Recovery PO three times daily (TID) until surgery. Within 2 days following surgery, patients may continue to receive Impact Advanced Recovery via feeding tube at the discretion of the treating physician.

After completion of study, patients are followed up at 24 and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Resectable, locally advanced esophageal cancer (adenocarcinoma, squamous cell, other histology).
* Medically operable.
* Treatment plan for (i) chemoradiation then surgery or chemotherapy followed by chemoradiation then surgery, or (ii) salvage esophagectomy.
* Able to tolerate feeds either orally or via tube gastrostomy or enterostomy.

Exclusion Criteria:

* Allergy to supplement.
* Pregnant.
* Hepatic insufficiency.
* Serum creatinine > 2.0.
* Metastatic disease.
* Performance status of > or equal to 2.
* Inability to take either oral intake or enteral feeds or both.
* Given increased rates of perioperative morbidity and mortality historically observed at our institution, patients undergoing salvage resection for squamous cell carcinoma will not be eligible for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Patient well-being improvement | Up to 30 days post-surgery
  Will be measured by weight loss change incurred during the course of therapy and maintenance of patient performance status. The composite outcome will be Clavien-Dindo postoperative morbidity (POM) score, which is an ordinal health quality outcome variable with six levels: 0=normal recovery, 1=minor complication, 2=complication requiring pharmaceutical intervention, 3=complication requiring surgical, endoscopic or radiological intervention, 4=life-threatening complication requiring intensive care and 5=complication leading to the patient's death. Each patient will be monitored for up to 30 days after their operation, and their POM score based on this postoperative period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L Hofstetter, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org